CLINICAL TRIAL: NCT03779555
Title: Lenalidomide Adherence in Older Adults: A Pilot Prospective Cohort Study of Oral Therapy for Multiple Myeloma
Brief Title: Lenalidomide Adherence in Older Adults
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left the university
Sponsor: Washington University School of Medicine (Other)
Collaborators: Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 201812141
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Micro-Electrical-Mechanical Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients taking lenalidomide for multiple myeloma: -Patients will be seen at baseline, 1 month (+/- 1 week), 2 months (3-5 weeks following 1-month assessment), and 3 months (3-5 weeks after 2-month follow-up)
  Interventions: Other: Medication Event Monitoring System

INTERVENTIONS:
Other: Medication Event Monitoring System — -Microchipped bottle cap
  Other Names: MEMS

SUMMARY:
To describe patterns of adherence and pilot baseline measures to investigate factors associated with lower adherence to lenalidomide in older adults with myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65
* Receiving lenalidomide for treatment of multiple myeloma.
* Anticipated to receive ongoing care at Siteman Cancer Center and its satellite sites
* Able to read and understand English.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Estimated life expectancy <6 months.
* Anticipated duration of lenalidomide therapy <3 months.
* Residing in a nursing facility where their medications are administered to them OR patient reports they do not self-administer their own medications.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants from Siteman Cancer Center and its satellite sites with multiple myeloma who are taking lenalidomide.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Adherence rate as measured by the number of days in which the lenalidomide pill bottle was open | Through completion of study (estimated to be 3 months)
  -Participants will be given a pill diary in which they will record if they opened the pill bottle without taking a medication (e.g. to ascertain remaining supply) to adjust the adherence rate accordingly

SECONDARY OUTCOMES:
Adherence rate as measured by a modified Brief Adherence Rating Scale | Through completion of study (estimated to be 3 months)
  * Participants will fill out a brief survey about taking lenalidomide and an estimate of their adherence using a visual analog scale
  * Scored 0-100%, 0% = lenalidomide not taken on any days and 100% = lenalidomide taken every day

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Fiala, MSW, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silberstein AE, Fiala MA, Loh KP, Cordner T, Mian H, Wildes TM. A pilot study of adherence to lenalidomide among older patients with multiple myeloma. J Geriatr Oncol. 2023 Sep;14(7):101560. doi: 10.1016/j.jgo.2023.101560. Epub 2023 Jun 27. No abstract available. PMID 37380519
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu